CLINICAL TRIAL: NCT01160367
Title: Trial of Ascertaining Individual Preferences for Loved One's Role in End-of-Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Chicago (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: NA_00010044; 5R01NR010733-02 (NIH)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Amyotrophic Lateral Sclerosis; GI Cancer; Pancreatic Cancer
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Gastrointestinal Neoplasms; Pancreatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard of care health decision making (Active Comparator): Patient-family dyads will receive the standard of care for support of patient and family members health care decision making during a clinic appointment.
  Interventions: Other: standard of care
- TAILORED intervention (Experimental): Patients and family members who receive the TAILORED Decision Making Intervention
  Interventions: Other: TAILORED Patient Family Decision Making

INTERVENTIONS:
Other: TAILORED Patient Family Decision Making — Patient-family dyads will receive TAILORED intervention on health decision making
  Arms: TAILORED intervention
Other: standard of care — Patient-family dyads will receive standard of care in health decision-making
  Arms: standard of care health decision making

SUMMARY:
Specific Aims and Hypotheses:

Aim 1: To test the effect of the "Trial of Ascertaining Individual preferences for Loved Ones' Role in End-of-life Decisions" (TAILORED) Intervention on family decision-making self-efficacy at 8 weeks both with respect to the patient's present situation and in a hypothetical situation in which the patient lacks decision-making capacity.

Hypotheses 1a: Family decision-making self-efficacy will be greater at 8 weeks in pairs that have undergone the TAILORED Intervention than in pairs receiving the standard information on advance directives in the patient's present situation.

Hypotheses 1b: Family decision-making self-efficacy will be greater at 8 weeks in pairs that have undergone the TAILORED Intervention than in pairs receiving the standard information on advance directives in the hypothetical situation in which the patient lacks decision making capacity.

Aim 2: To test the effect of the TAILORED Intervention on family psychological outcomes (depression, caregiver burden, decision making distress).

Hypotheses 2a: Depression will be less at 8 weeks in family members who have undergone the TAILORED Intervention than in family members who have received the standard information on advance directives.

Hypotheses 2b: Caregiver burden will be less at 8 weeks in family members who have undergone the TAILORED Intervention than in family members who have received the standard information on advance directives.

Hypotheses 2c: Decision-making distress will be less at 8 weeks in family members who have undergone the TAILORED Intervention than in family members who have received the standard information on advance directives.

Aim 3: To test the effect of the TAILORED Intervention on patient and family satisfaction with family decision-making involvement.

Hypothesis 3a: Patient satisfaction with family decision involvement will be greater at 8 weeks in patients who have undergone the TAILORED Intervention than in patients receiving the standard information on advance directives.

Hypothesis 3b: Family member satisfaction with decision involvement will be greater at 8 weeks in family members who have undergone the TAILORED Intervention than in family members receiving the standard information on advance directives.

Aim 4: To explore family decision-making self-efficacy and perceptions of the TAILORED Intervention.

DETAILED DESCRIPTION:
Enhanced patient-family health care decision making is essential to improving the overall quality of end-of-life care (NIH State of the Science Conference Statement on Improving End-of-Life Care, 2004). Although most terminally ill patients desire shared family decision making, few family members are prepared for this and many report high levels of distress, and even the inability to make such decisions (Nolan, et al., 2005). Factors positively influencing the surrogates are: 1) previous experience with surrogate decision making, 2) knowing the patient's preferences, and 3) receiving positive reinforcement about decision making. The last two are amenable to change in "Trial of Ascertaining Individual preferences for Loved Ones' Role in End-of-life Decisions" (the "TAILORED" study). The TAILORED intervention is a simple clinic- based protocol involving an assessment of the confidence (self-efficacy) of family members for making health care decisions with or for a terminally ill loved one. Clinicians then tailor their guidance to patients and families about issues to discuss at home to better prepare family members for the desired decision-making role. This randomized clinical trial will include 132 patient-family dyads from two diagnostic groups: a group expected to retain (amyotrophic lateral sclerosis) or lose decisional capacity (advanced gastro-intestinal malignancy). A nurse will deliver the TAILORED intervention in the clinic at baseline and will call the family member in 4- weeks to encourage ongoing patient-family discussion. Outcomes will be assessed at 8-weeks. A subgroup of family members whose loved one has died will be interviewed in-depth about their end-of-life decision making and the impact of the TAILORED Intervention. Aim 1: To test the effect of the TAILORED intervention on family decision-making self-efficacy at 8 weeks both with respect to the patient's present situation and in a hypothetical situation in which the patient lacks decision-making capacity. Aim 2: To test the effect of the TAILORED intervention on family psychological outcomes (depression, caregiver burden, decision making distress). Aim 3: To test the effect of the TAILORED intervention on patient and family satisfaction with family decision-making involvement. Aim 4: To explore family decision-making self-efficacy and perceptions of the TAILORED intervention. PUBLIC HEALTH RELEVANCE: Although most terminally ill patients prefer to share health care decision making with family and want family to make decisions for them if they are too ill to do so, few family members are prepared for this role and many report high levels of distress and even the inability to make such decisions. "Trial of Ascertaining Individual preferences for Loved Ones' Role in End-of-life Decisions" (the "TAILORED" study) tests a simple clinic-based protocol that allows clinicians to assess the confidence (self-efficacy) of family members for making health care decisions with or for a terminally ill loved one. Clinicians then tailor their guidance to patients and families about what issues to discuss to better prepare family members for the decision making role desired by the patient.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria

1. Age 18 or older
2. Speaks and reads English
3. Diagnosed by a specialist at either Johns Hopkins Medical Institutions or University of Chicago Medical Center as having ALS or stage III or IV GI or pancreatic cancer.
4. Accompanied to clinic by a family member who may participate in the patient's health care decisions and who patient gives permission to approach for participation in study.
5. Lives within a 2-hour drive of The Johns Hopkins Medical Institutions or The University of Chicago Medical Center

5.G.2. Family Inclusion Criteria

1. Age 18 or older
2. Speaks and reads English
3. Identified by the patient-subject as a family member whom the patient may involve in health care decision making in the present and/or should the patient become too ill to make health care decisions.
4. Person who the patient-subject has granted investigators permission to approach for participation in this study.

Exclusion Criteria:

* Patient Exclusion Criteria

  1. Severe visual impairment that would limit ability to visualize instrument illustrations
  2. Cognitive impairment indicated by a Short Portable Mental Status Questionnaire adjusted error score of >5
  3. Has no family member who might assist in decision making or family member declines to participate.
  4. Is not accompanied to the clinic by family member.
  5. G.4. Family Exclusion Criteria

  <!-- -->

  1. Declines to participate.
  2. Severe visual impairment that would limit ability to visualize instrument illustrations.
  3. Cognitive impairment indicated by a Short Portable Mental Status Questionnaire adjusted error score of >5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2010-08-26 (Actual); Primary Completion 2014-03-26 (Actual); Study Completion 2014-03-26 (Actual)

PRIMARY OUTCOMES:
family decision-making self-efficacy | at 8 weeks after the intervention

SECONDARY OUTCOMES:
family psychological outcomes (depression, caregiver burden, decision making distress) | 8 weeks after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sulmasy DP, Hughes MT, Yenokyan G, Kub J, Terry PB, Astrow AB, Johnson JA, Ho G, Nolan MT. The Trial of Ascertaining Individual Preferences for Loved Ones' Role in End-of-Life Decisions (TAILORED) Study: A Randomized Controlled Trial to Improve Surrogate Decision Making. J Pain Symptom Manage. 2017 Oct;54(4):455-465. doi: 10.1016/j.jpainsymman.2017.07.004. Epub 2017 Jul 14. PMID 28712987